CLINICAL TRIAL: NCT05582876
Title: Multicenter Assessment of Clinical Utility PET / MR With the Use of the Radiotracer 68Ga-PSMA-11 in Therapy Planning Personalized in Patients With Prostate Cancer
Acronym: PROSPETMR2021
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/ABM/01/00074
Record Dates: First submitted 2022-10-11; First posted 2022-10-17 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: PET/CT; PET/MR; 68Ga-PSMA-11; PSA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1- patient of middle and high risk of prostate cancer (Active Comparator): Patients with diagnosis or high probability of prostate cancer medium and high risk according to ISUP for which implementation is planned radical treatment [i.e. PSA≥10 ng / ml or GS ≥ 7 (ISUP ≥2) or ≥cT2b].
  Interventions: Radiation: Radiopharmaceutical 68Ga-PSMA-11 PET/CT
- Group 2- patient after radical treatment, at relapse biochemical (Active Comparator): Prostate cancer patients after radical treatment, with recurrence biochemical tests according to the criteria of the European Society of Urology (EAU, European Association of Urology) [at least double measurement PSA ≥0.2 ng / ml not earlier than 6-13 weeks after radical prostatectomy or PSA≥0.1 with PSAdt (PSA doubling time) <3 months or increase in PSA after radical radiotherapy> 2 ng / ml above PSAnadir - the lowest PSA value found after the test treatment] for whom further treatment is planned and the test result imaging / molecular imaging may alter the therapeutic decision
  Interventions: Radiation: Radiopharmaceutical 68Ga-PSMA-11 PET/CT

INTERVENTIONS:
Radiation: Radiopharmaceutical 68Ga-PSMA-11 PET/CT — The radiopharmaceutical will be administered intravenously in doses with an activity of 1.8-2.2 MBq / kg b.w.

SUMMARY:
The aim of multicentre phase 3 trial is evidence diagnostic value of 68Ga-PSMA-11 (in PET / CT and PET / MR techniques) in patients with high-risk and intermediate prostate cancer before radical treatment and in diagnosed patients biochemical recurrence after radical treatment

ELIGIBILITY:
Inclusion Criteria:

Group 1. Patients with diagnosis or high probability of medium and high prostate cancer according International Society of Urological Pathology (ISUP) risk for whom radical treatment is planned

* Prostate adenocarcinoma confirmed by biopsy and histopathological examination
* Results indicating a moderate RGK (Gleason score 7 or cT2b or PSA 10-20 ng / ml) or high (Gleason score> 7 or cT2c or PSA> 20 ng / ml) risk according to ISUP
* Creatinine value allowing for safe PET / MR examination with a contrast agent: creatinine less than or equal to 1.5 times the upper limit of normal, creatinine clearance> 60 mL / min
* Age ≥18 years
* Signing informed consent to participate in the study
* Pelvic / prostate mpMR examination performed, not earlier than 30 days before inclusion in the study

Group 2. Patients with RGK after radical treatment, with biochemical recurrence according to EAU criteria, who are scheduled for further treatment and the result of the imaging / molecular examination may affect change of therapeutic decision:

* Prostate adenocarcinoma confirmed by biopsy and histopathological examination
* After radical treatment
* In patients after radical prostatectomy: with at least two PSA measurements ≥0.2 ng / ml not earlier than after 6-13 weeks after radical prostatectomy or PSA≥0.1 with PSAdt (PSA doubling time) <3 months PSA on at least two consecutive studies in consecutive last 6 months before qualification (last determination within 6 weeks before qualification) Or
* In patients after radical radiotherapy: biochemical recurrence defined as nadir PSA + 2 ng / ml
* Age ≥18 years
* Signing informed consent

Exclusion Criteria:

* Presence of metallic foreign bodies / implants / prostheses / stimulators etc. inside the body, the possession of which is a contraindication to the MR 3T examination
* Claustrophobia
* Patient size precluding PET / MR examination due to diameter gantry
* Known contraindications for the use of radiopharmaceuticals or substances auxiliary (e.g. renal failure and allergy to ingredients in the preparation)
* Treatment for malignant neoplasm not associated with the prostate gland
* Participating in another clinical trial
* Lack of informed consent to participate in the study
* Age <18 years

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Sensivity of the radiopharmaceutical 68Ga-PSMA-11 compared to PET/MR and PET/CT | 24 months
  Validation of the diagnostic value of 68Ga-PSMA-11 (in PET / CT and PET / MR techniques) in the assessment stage of prostate cancer and precise assessment of the location of neoplastic changes.

SECONDARY OUTCOMES:
Establishing a therapeutic path depending on the PET/MR and PET/CT | 24 months
  Percentage of patients with 68Ga-PSMA-11 PET / CT and 68Ga-PSMA-11 PET / MR will lead to a change in the therapeutic path
Detection of the site of recurrence | 24 months
  Comparison of the frequency of detecting the site of recurrence after examination with standard methods, 68Ga-PSMA-11 PET / CT and 68Ga-PSMA-11 PET / MR (only for the second group)
Determination of PSA concentration | 24 months
  Determination of the PSA concentration at which the 68Ga-PSMA-11 PET / MR test enables detection of local or regional recurrence (only for the second group)
Number of participants with adverse events related to 68Ga-PSMA-11 | 24 months
  Serious adverse events are not expected. The radiotracer 68Ga-PSMA-11 is dose by the intravenous route in trace amounts and does not affect the patient's well-being.
  The use of 68Ga-PSMA-11 is contraindicated in kidney failure and allergies to the ingredients of the preparation (all patients will have their serum creatinine measured before the test).
Absorbed radiation dose | 24 months
  Assessment and comparison of the absorbed radiation dose during the 68Ga-PSMA-11 PET / CT examination and 68Ga-PSMA-11 PET / MR
Evaluation of pharmacoeconomic data | 24 months
  Comparison of the costs of the procedures planned for performance after the first visit, and those that were actually made after conducting the assessed tests

CONTACTS AND LOCATIONS:
Locations (7):
- Poland (7):
  - Białystok Oncology Center Maria Skłodowska-Curie, Bialystok
  - University Clinical Hospital in Białystok, Bialystok
  - Independent Public Health Care Center of the Ministry of Internal Affairs and Administration in Białystok, Bialystok
  - Laboratory of Molecular Imaging and Technology Development, Bialystok
  - Oncology Center named after prof. F. Łukaszczyk in Bydgoszcz, Bydgoszcz
  - Provincial Multidisciplinary Center of Oncology and Traumatology named after M. Copernicus University in Łódź, Lodz
  - Center of Oncology of the Lublin Region St. Jana z Dukli, Lublin